CLINICAL TRIAL: NCT05592054
Title: PROximal TEmporary oCclusion Using Balloon Guide Catheter for Mechanical Thrombectomy(PROTECT-MT)
Brief Title: Proximal TEmporary oCclusion Using Balloon Guide Catheter for Mechanical Thrombectomy
Acronym: PROTECT-MT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB suggestion
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jian-min Liu, Director of Cerebrovascular Disease Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROTECT-MT
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Thrombectomy; Thrombosis
MeSH Terms: conditions — Ischemic Stroke; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Balloon guide catheters (BGCs)
  Interventions: Procedure: Balloon guide catheters (BGCs)
- Control group (Active Comparator): Standard guide catheter
  Interventions: Procedure: Standard guide catheter

INTERVENTIONS:
Procedure: Balloon guide catheters (BGCs) — MT procedure with Balloon guide catheters (BGCs)
  Arms: Intervention group
Procedure: Standard guide catheter — MT procedure with standard guide catheter
  Arms: Control group

SUMMARY:
A multi-center, prospective, randomized, open-label, blinded endpoint assessment (PROBE) clinical trial of endovascular treatment among selected AIS.

DETAILED DESCRIPTION:
The PROTECT-MT study is a prospective, multicenter, randomized controlled, open-label, blinded endpoint evaluation (PROBE) trial, and aims to determine the effectiveness of balloon guide catheter(BGC) as compared to standard guide catheter on functional outcome (modified Rankin Scale [mRS] score at Day 90) in patients with acute ischemic stroke due to anterior circulation large vessel occlusion.

Primary Endpoints

Functional outcome, defined as modified Rankin Scale (mRS) score, at 90 days (±14 days) .

Secondary Endpoints

1. Dichotomized mRS at 90 days after the operation (0-1 versus 2-6, 0-2 versus 3-6, 0-3 versus 4-6, 0-4 versus 5-6, 0-5 versus 6).
2. Change in stroke severity (NIHSS score) at 24 hours post treatment.
3. Change in stroke severity (NIHSS score) at 7 days post treatment or discharge (whichever occurs first).
4. Final infarct volume at 5-7 days post treatment
5. Technical success rate (defined as successfully navigating the guide catheter into the target vessel, and finishing the mechanical thrombectomy procedure without changing to another guide catheter).
6. Reperfusion outcome (eTICI 2b or greater, eTICI 2c or greater, eTICI 3) in final angiogram.
7. Reperfusion outcome (eTICI 2b or greater, eTICI 2c or greater, eTICI 3) after the first pass.
8. Time from groin puncture to successful reperfusion (eTICI 2b or greater, eTICI 2c or greater).
9. Percentage of subjects with acceptable revascularization quality (eTICI 2b or greater, eTICI 2c or greater) within 45 min of access.
10. Number of thrombectomy attempts (final).
11. Occurrence of emboli to a new territory.

Safety Endpoints:

1. Deaths at 90 days (±14 days) post treatment.
2. Intracranial hemorrhage, symptomatic intracranial hemorrhage or asymptomatic intracranial hemorrhage at 7 days post treatment or discharge (whichever occurs first).
3. Other serious adverse events (SAEs) adjudicated by the Clinical Events Committee.
4. Any Procedural complications, including vessel dissection, arterial perforation, and femoral access complications, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of AIS with confirmed anterior circulation LVO (including intracranial segment of the internal carotid artery, and the first or proximal second segment [M1 or proximal M2] of the middle cerebral artery) by brain imaging
3. To receive MT within 24 hours after AIS onset according to local guidelines
4. Preoperative mRS score of 0-1
5. Signed informed consent form obtained from the subject (or approved surrogate)

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by imaging
2. Known or suspected pre-existing (chronic) large vessel occlusion in the symptomatic territory
3. Excessive vascular access tortuosity disables the use of balloon guide catheter
4. Intracranial stent implanted in the same vascular territory that precludes the safe deployment/removal of the neuro-thrombectomy device
5. Any other condition that precludes the performing of mechanical thrombectomy procedure
6. Occlusions in multiple vascular territories confirmed by Computed Tomography Angiography(CTA) or Magnetic Resonance Angiography(MRA)
7. Subjects who are pregnant
8. Subjects who are allergy to the contrast agent
9. Subjects who refuse to cooperate or unable to tolerate interventional operation
10. Subjects whose expected lifetime are less than 90 days
11. Subjects who are unlikely to participate in follow-up assessments according to the investigator's judgement
12. Any other condition that, according to the investigator's judgement, not suitable for using of balloon guide catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 90 days
  defined as modified Rankin Scale (mRS) score shift

SECONDARY OUTCOMES:
Dichotomized mRS | 90 days
  Dichotomized mRS (0-1 versus 2-6,0-2 versus 3-6,0-3 versus 4-6,0-4 versus 5-6,0-5 versus 6)
Change in stroke severity | 24 hours post treatment
  NIHSS
Change in stroke severity | 7 days post treatment or discharge (whichever occurs first).
  NIHSS
Final infarct volume | 5-7 days post treatment
  Final infarct volume at 5-7 days post treatment
Technical success rate | 24 hours after mechanical thrombectomy
  defined as successfully navigating the guide catheter into the target vessel, and finishing the mechanical thrombectomy procedure without changing to another guide catheter
Reperfusion outcome | 24 hours after mechanical thrombectomy
  (eTICI 2b or greater ,eTICI 2c or greater, eTICI 3)in Final angiogram.
Reperfusion outcome | 24 hours after mechanical thrombectomy
  (eTICI 2b or greater ,eTICI 2c or greater, eTICI 3) after First pass
Time from groin puncture to successful reperfusion | 24 hours after mechanical thrombectomy
  eTICI 2b or greater, eTICI 2c or greater
Revascularization quality | 24 hours after mechanical thrombectomy
  Percentage of subjects with acceptable revascularization quality (eTICI 2b or greater, eTICI 2c or greater) within 45 min of access
Thrombectomy attempt (final) | 24 hours after mechanical thrombectomy
  Number of thrombectomy attempts (final)
Occurrence of emboli to a new territory | 24 hours after mechanical thrombectomy
  Occurrence of emboli to a new territory

OTHER OUTCOMES:
Death | 90 days
  Deaths at 90 days (±14 days) post treatment
Intracerebral hemorrhage (ICH) | 7 days post treatment or discharge (whichever occurs first)
  Intracranial hemorrhage, symptomatic intracranial hemorrhage or asymptomatic intracranial hemorrhage at 7 days post treatment or discharge (whichever occurs first)
SAE | 90 days
  Other serious adverse events (SAEs) adjudicated by the Clinical Events Committee
perioperative complications | Perioperative period
  Any peri-procedural complications, including vessel dissection, arterial perforation, and femoral access complications, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Jianimin Liu, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to Oriental Collaboration group on Emerging Advanced therapy for Neurovascular diseases Consortium.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: http://www.ocin.org.cn/about

REFERENCES:
- [Derived] Liu J, Zhou Y, Zhang L, Li Z, Chen W, Zhu Y, Yao X, Zhang L, Liu S, Peng Y, Wei M, Zhang Q, Shu H, Wang S, Liu W, Wan S, Li T, Fang Y, Han H, Zhang G, Huang L, Wang F, Cheng G, Gao L, Shi H, Han J, Luo Y, Li S, Cai C, Yin R, Jin Z, Shao C, Tian B, Zhang Y, Li Q, Zhang Y, Zhang P, Li B, Xing P, Shen H, Zhu X, Zhang X, Hua W, Shen F, Huyan M, Chen R, Zuo Q, Li Q, Huang Q, Xu Y, Deng B, Zhao R, Goyal M, Zhang Y, Yang P; PROTECT-MT Investigators. Balloon guide catheters for endovascular thrombectomy in patients with acute ischaemic stroke due to large-vessel occlusion in China (PROTECT-MT): a multicentre, open-label, blinded-endpoint, randomised controlled trial. Lancet. 2024 Nov 30;404(10468):2165-2174. doi: 10.1016/S0140-6736(24)02315-8. Epub 2024 Nov 20. PMID 39579782

DOCUMENTS (2):
  • Study Protocol (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT05592054/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT05592054/SAP_001.pdf